CLINICAL TRIAL: NCT05338437
Title: Neuromuscular Electrical Stimulation in Heart Failure Patients to Improve Functional Recovery Following Hospitalization (NeuHF-Recover)
Brief Title: NMES in HF Patients to Improve Functional Recovery Following Hospitalization
Acronym: NeuHFRecover
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Sherrie Khadanga, Associate Director Cardiac Rehabilitation, University of Vermont Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00001757
Record Dates: First submitted 2022-03-21; First posted 2022-04-21 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: HF, rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Neuromuscular electrical stimulation (Experimental): Neuromuscular electrical stimulation of the quadriceps. 45 minutes, 5 days per week
  Interventions: Device: Neuromuscular electrical stimulation
- Control (No Intervention): No treatment control

INTERVENTIONS:
Device: Neuromuscular electrical stimulation — Bilateral quadriceps muscle stimulation
  Arms: Neuromuscular electrical stimulation

SUMMARY:
The goal of this research study is to understand whether an at-home exercise program started after hospitalization for HFpEF, and continuing for 4 weeks following discharge from the hospital, can preserve or improve physical function.

DETAILED DESCRIPTION:
Heart failure is the leading cause of hospitalization among adults in the US with patients with preserved ejection fraction (HFpEF) comprising half of those admissions. Many patients exhibit chronic fatigue, exercise intolerance and an inability to perform activities of daily living, which is exacerbated by hospitalization. The goal of this research study is to understand whether an at-home exercise program started soon after hospitalization and continuing for 4 weeks following discharge can improve functional recovery in HFpEF patients. Volunteers will be randomly assigned to receive neuromuscular electrical stimulation (NMES) of their quadriceps muscles or not to receive NMES (control group). Volunteers will be evaluated during hospitalization and 4 weeks following discharge. Assessments will include measurements of physical function by 6 minute walk test and the Short Physical Performance Battery, as well as assessment of subjective physical functional capacity and quality of life using the Medical Outcomes Short form 36 and Kansas City Cardiomyopathy questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 50-90 years of age
* clinical diagnosis of HF being actively managed during hospitalization
* live within 30 miles of the medical center
* able to perform informed consent

Exclusion Criteria:

* rheumatoid arthritis or other inflammatory/autoimmune disease
* cancer, excluding non-melanoma skin cancer or low-grade prostate cancer
* severe dementia/alzheimer's disease
* exercise limiting peripheral vascular disease
* neuromuscular disease or neuromuscular dysfunction associated with cerebrovascular event
* body mass index ≥40 kg/m2
* lower extremity blood clot or implantable cardioverter-defibrillator or pacemaker

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Distance (6MW) | Change from Hospital Discharge (Within 1 day) to 4-weeks post-discharge
  6 MW was developed to assess cardiopulmonary fitness in patients with lung and cardiac disease, and has been validated in heart failure patients. It assesses the distance that a patient can walk in 6 minutes time around a standard course.

SECONDARY OUTCOMES:
Short Physical Performance Battery | Change from Hospital Discharge (Within 1 day) to 4-weeks post-discharge
  Short Physical Performance Battery is composed of three tasks assessing balance, gait speed, and ability to stand from a chair. Units on a scale for each domain range from of 0-4 for a total score of 0 to 12, with a higher score indicating better physical function.
Medical Outcomes Short Form 36 | Hospital discharge (Within 1 day) and 4-weeks post-discharge
  The Medical Outcomes Short Form 36 is a questionnaire that assesses self-reported health and physical functional status. There are 36 questions that reflect eight sub-domains of health included in this questionnaire. Scores for each domain represent weighted sums of the questions in each sub-domain. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. This measure represents the total computed score across all sub-domains. Lower scores represent worse overall health, while higher scores represent better health.
Medical Outcomes Short Form 36 - Role Emotional | Hospital discharge (Within 1 day) and 4-weeks post-discharge
  The Medical Outcomes Short Form 36 is a questionnaire that assesses self-reported health and physical functional status. There are 36 questions that reflect eight sub-domains of health included in this questionnaire. Scores for each domain represent weighted sums of the questions in each sub-domain. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. This sub-domain focuses on limitations in usual role activities because of emotional problems. Lower scores represent more limitations, while higher scores represent less limitations.
Medical Outcomes Short Form 36 - Social Function | Hospital discharge (Within 1 day) and 4-weeks post-discharge
  The Medical Outcomes Short Form 36 is a questionnaire that assesses self-reported health and physical functional status. There are 36 questions that reflect eight sub-domains of health included in this questionnaire. Scores for each domain represent weighted sums of the questions in each sub-domain. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. This sub-domain focuses on limitations in social activities because of physical or emotional problems. Lower scores represent more more limitations, while higher scores represent less limitations.
Medical Outcomes Short Form 36 - Vitality | Hospital discharge (Within 1 day) and 4-weeks post-discharge
  The Medical Outcomes Short Form 36 is a questionnaire that assesses self-reported health and physical functional status. There are 36 questions that reflect eight sub-domains of health included in this questionnaire. Scores for each domain represent weighted sums of the questions in each sub-domain. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. This sub-domain focused on vitality (energy and fatigue). Lower scores represent less vitality, while higher scores represent more vitality.
Medical Outcomes Short Form 36 - General Health | Hospital discharge (Within 1 day) and 4-weeks post-discharge
  The Medical Outcomes Short Form 36 is a questionnaire that assesses self-reported health and physical functional status. There are 36 questions that reflect eight sub-domains of health included in this questionnaire. Scores for each domain represent weighted sums of the questions in each sub-domain. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. This sub-domain focused on self-reported general health. Lower scores represent worse health, while higher scores represent better health.
Medical Outcomes Short Form 36 - Bodily Pain | Hospital discharge (Within 1 day) and 4-weeks post-discharge
  The Medical Outcomes Short Form 36 is a questionnaire that assesses self-reported health and physical functional status. There are 36 questions that reflect eight sub-domains of health included in this questionnaire. Scores for each domain represent weighted sums of the questions in each sub-domain. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. This sub-domain focused on self-reported general health. Lower scores represent worse health, while higher scores represent better health.
Medical Outcome Short Form 36 - Role Physical | Hospital discharge (Within 1 day) and 4-weeks post-discharge
  The Medical Outcomes Short Form 36 is a questionnaire that assesses self-reported health and physical functional status. There are 36 questions that reflect eight sub-domains of health included in this questionnaire. Scores for each domain represent weighted sums of the questions in each sub-domain. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. This sub-domain focused on self-reported general health. Lower scores represent worse health, while higher scores represent better health.
Medical Outcomes Short Form 36 - Physical Function | Hospital discharge (Within 1 day) and 4-weeks post-discharge
  The Medical Outcomes Short Form 36 is a questionnaire that assesses self-reported health and physical functional status. There are 36 questions that reflect eight sub-domains of health included in this questionnaire. Scores for each domain represent weighted sums of the questions in each sub-domain. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. This sub-domain focused on self-reported general health. Lower scores represent worse health, while higher scores represent better health.
Katz Index of Independence in Activities of Daily Living | Hospital discharge (Within 1 day) and 4-weeks post-discharge
  The Katz Index of Independence in Activities of Daily Living, commonly referred to as the Katz ADL, is the most appropriate instrument to assess functional status as a measurement of the client's ability to perform activities of daily living independently. Clinicians typically use the tool to detect problems in performing activities of daily living and to plan care accordingly. The Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. Clients are scored yes/no for independence in each of the six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
Lawton Instrumental Activities of Daily Living (IADL) Scale | Hospital discharge (Within 1 day) and 4-weeks post-discharge
  The Lawton Instrumental Activities of Daily Living Scale (IADL) is an appropriate instrument to assess independent living skills. These skills are considered more complex than the basic activities of daily living as measured by the Katz Index of ADLs. The instrument is most useful for identifying how a person is functioning at the present time, and to identify improvement or deterioration over time. There are eight domains of function measured with the Lawton IADL scale. Women are scored on all 8 areas of function; historically, for men, the areas of food preparation, housekeeping, laundering are excluded.
  Clients are scored according to their highest level of functioning in that category. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT05338437/Prot_SAP_001.pdf